CLINICAL TRIAL: NCT05602532
Title: Triglyceride-Glucose Index in Diabetic Nephropathy in Type 2diaberes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abo Elyosr Garhey Yonis, Doctor, Assiut University
Other Study IDs: TYG index in DN in type 2 DM
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to investigate the associations between the TyG index and diabetic nephropathy in patients with type2 DM .

DETAILED DESCRIPTION:
the triglyceride-glucose (TyG) index was proposed as a simple and reliable surrogate marker of IR, and it has been reported to be closely correlated with the HOMA-IR index. The TyG index has the advantage of being applicable in clinical practice since both triglyceride and glucose levels are routinely measured and the cost of these measurements is low.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 DM

Exclusion Criteria:

- (1) Individuals with obstructive uropathy, severe heart failure, stroke, liver disease, cancer, autoimmune disease (2) Pregnant woman. (3)End stage renal disease patients on dialysis ( glomerular filtration rate <15 mL/min/1.73 m2) or renal transplantation.

(4) Type 1 Diabetic patient. (5) Albuminuria due to non-diabetic renal disease

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There will be no risk for the patients during the study Confidentiality will be assured. The participants will be informed about the research and they will hsve the right to refuse to participate.
  Written consents will be obtained from all the participants; illiterate participants will give their consent by fingerprints.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
TyG index in type 2diaberes Mellitus | Baseline
  Detecting the association between the TyG index and diabetic nephropathy in type 2 diabetes

REFERENCES:
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Beckman JA, Creager MA, Libby P. Diabetes and atherosclerosis: epidemiology, pathophysiology, and management. JAMA. 2002 May 15;287(19):2570-81. doi: 10.1001/jama.287.19.2570. PMID 12020339
- [Background] Yamagishi S, Imaizumi T. Diabetic vascular complications: pathophysiology, biochemical basis and potential therapeutic strategy. Curr Pharm Des. 2005;11(18):2279-99. doi: 10.2174/1381612054367300. PMID 16022668
- [Background] Liang S, Cai GY, Chen XM. Clinical and pathological factors associated with progression of diabetic nephropathy. Nephrology (Carlton). 2017 Dec;22 Suppl 4:14-19. doi: 10.1111/nep.13182. PMID 29155497
- [Background] Lee MY, Hsiao PJ, Huang JC, Hsu WH, Chen SC, Chang JM, Shin SJ. ASSOCIATIONS BETWEEN TRIGLYCERIDE/HIGH-DENSITY LIPOPROTEIN CHOLESTEROL RATIO AND MICRO- AND MACROANGIOPATHIES IN TYPE 2 DIABETES MELLITUS. Endocr Pract. 2018 Jul;24(7):615-621. doi: 10.4158/EP-2017-0254. PMID 30048164